CLINICAL TRIAL: NCT06721039
Title: Comparison of Ultrasound-Guided Quadratus Lumborum Plane Block Versus Intraperitoneal and Periportal Bupivacaine Infiltration in Postoperative Analgesia After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: medina medical center (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Salah Elsawy, lecturere of anaesthesia and intensive care, medina medical center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS 168/2022
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2022-03

CONDITIONS: Quadratus Lumborum; Laparoscopic Cholecystectomy; Ultrasound Guided; Post Operative Analgesia
Keywords: Quadratus Lumborum Plane Block, Intraperitoneal and Periportal Bupivacaine Infiltration, Post Operative Analgesia, Laparoscopic Cholecystectomy
MeSH Terms: interventions — Infusions, Parenteral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Bilateral QL block: sonovisible block needle will be inserted under ultra-sonographic monitoring between the iliac wing and rib at the midaxillary line for the TQL block in the lateral decubitus positioning of the patient. The space between the quadratus lumborum and psoas major muscles will be visualized with Ultrasound Guided and 0.25% bupivacaine will be injected after visualization of the tip of the needle reaching the plane, 2ml of anaesthetic solution will be instilled to view the hydro dissection, confirming the correct placement. Following this, the total volume of 40 ml of 0.25% bupivacaine will be instilled, creating a meniscus between the planes
  Interventions: Drug: Bilateral QL block
- Group 2 (Active Comparator): Intraperitoneal and port sites infiltration with 40 ml of 0.25% bupivacaine will be injected under the direct vision into the hepato-diaphragmatic space, near and above the hepato-duodenal ligament and above the gall bladder also injected at the port sites at the end of operation before removal of the probes
  Interventions: Drug: Intraperitoneal and port sites infiltration

INTERVENTIONS:
Drug: Bilateral QL block — sonovisible block needle will be inserted under ultra-sonographic monitoring between the iliac wing and rib at the midaxillary line for the TQL block in the lateral decubitus positioning of the patient. The space between the quadratus lumborum and psoas major muscles will be visualized with Ultrasound Guided and 0.25% bupivacaine will be injected after visualization of the tip of the needle reaching the plane, 2ml of anaesthetic solution will be instilled to view the hydro dissection, confirming the correct placement. Following this, the total volume of 40 ml of 0.25% bupivacaine will be instilled, creating a meniscus between the planes
  Arms: Group 1
Drug: Intraperitoneal and port sites infiltration — with 40 ml of 0.25% bupivacaine will be injected under the direct vision into the hepato-diaphragmatic space, near and above the hepato-duodenal ligament and above the gall bladder also injected at the port sites at the end of operation before removal of the probes
  Arms: Group 2

SUMMARY:
The primary outcome: is measured by pain at rest and upon mobilization according to VAS. VAS for pain (ranging from 0 to 10, where 0 no pain and 10 maximum pain) will be evaluated postoperatively and every 2 hours during the first 6 hours and then every 6 hours for 24 hours postoperatively.

DETAILED DESCRIPTION:
Since the concept of day case surgeries is getting more popular, surgeons and anesthesiologists are trying their best to provide adequate post-operative analgesia. The proper management of post-operative pain ensures early ambulation of patients and obviates many post-operative complications.

The most common modality for post-operative pain management has remained the parenteral use of non-steroidal anti-inflammatory drugs (NSAIDs) and opioids.

Intraperitoneal and periportal infiltration with local anesthetic agents has also remained a popular method to take care of immediate postoperative pain. This technique is virtually cost-free, rapid, and hardly requires any special technical experience or equipment for its use. But as there are advances in anesthetic techniques, more and more regional blocks are being tried to take care of post-operative pain. The choice of anaesthetic block technique depends upon the site of surgical incision proposed.

Quadratus lumborum (QL) block is a posterior abdominal wall block which permits the spread of local anesthetic agent behind the quadratus lumborum muscle into a triangular space known as a lumbar interfacial triangle, which lies beside the middle layer of the thoracolumbar fascia.

This interfacial plane is in adjoining proximity with numerous sympathetic fibers and conjoin with the thoracic paravertebral space, thus preceding to a long-standing block with the capability to provide visceral analgesia (Kadam, 2013).

ELIGIBILITY:
Inclusion Criteria:

* Age 21-60 years of both sexes.
* Elective laparoscopic cholecystectomy under general anesthesia.
* Physical Status: ASA I and II patients after taking written and informed consent.

Exclusion Criteria:

* • Refusal of procedure or participation in the study by patients.

  * Physical status: ASA III or above.
  * Infection at site of injection.
  * Psychiatric illness that leads to inability to cooperate, speak or read.
  * Daily use of opioids.
  * History or evidence of coagulopathy especially if INR>1.5 and platelet <100.000
  * Allergies to drugs used (Bupivacaine 0.5%).

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-04-03 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
pain score postoperative | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University Faculty of Medicine, New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.